CLINICAL TRIAL: NCT04945148
Title: Oxidative Phosphorylation Targeting In Malignant Glioma Using Metformin Plus Radiotherapy Temozolomide
Acronym: OPTIMUM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hopital Foch (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019_0007
Record Dates: First submitted 2021-06-25; First posted 2021-06-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Glioblastoma, IDH-wildtype
Keywords: Glioblastoma; FGFR3-TACC3; Metformin; Radio-chemotherapy; OXPHOS+
MeSH Terms: conditions — Glioblastoma | interventions — Metformin; Radiation; Temozolomide

STUDY DESIGN:
Intervention Model Description: Metformin (1500 to 3000mg/day) in addition to Stupp protocol, starting 7 days before the start of the standard radiotherapy (RT, 60Gy/6 weeks), concomitant Temozolomide (TMZ) chemotherapy (75mg/m²/day), and adjuvant TMZ (150-200 mg/m2/ 5 days) + metformin will follow onwards until the 12th cycle of TMZ
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metformin (Experimental): Patients who have been selected with an OXPHOS+ status, will start standard radiotherapy (RT, 60Gy/6 weeks), concomitant TMZ chemotherapy (75mg/m²/day), and metformin by 7 weeks after surgery and adjuvant TMZ + metformin will follow onwards until the 12th cycle of TMZ. Patients still in remission after this time-point will continue metformin alone until progression.
  Interventions: Drug: Metformin; Radiation: Radiation IMRT; Drug: Temozolomide

INTERVENTIONS:
Drug: Metformin — Metformin 2000 to 3000mg/day daily will be started by 6 weeks after histological diagnosis and 7 days before the start of RT-TMZ and will continue until progression.
Radiation: Radiation IMRT — 2 Gy x 5 days for 6 weeks to be started 7 days after first administration of Metformin and by 7 weeks after histological diagnosis
  Other Names: Radiation
Drug: Temozolomide — 75 mg/m² daily from first to last day of radiation (IMRT) and then 150 to 200 mg/m² x 5 days every 28 days cycle for 12 cycles

SUMMARY:
Tailored approaches targeting crucial oncogenes and pathways have shown successful results in a number of cancer types and offer exciting perspective in neuro-oncology. IDH (Isocitrate dehydrogenase) wild-type (IDHwt) glioblastoma (GBM) (10%) present a unique and homogenous energetic metabolism which is specifically dependent on the oxidative phosphorylation (OXPHOS) rather than on the aerobic glycolysis. OXPHOS+ IDHwt GBMs overexpress mitochondrial markers and can be specifically inhibited by mitochondrial inhibitors in vitro and in vivo.

Metformin is an oral inhibitor of mitochondrial complex I and is a widely used drug in diabetic and non-diabetic patients, safe and well tolerated in association with radiotherapy and chemotherapy.

Basing on drastic effect, the investigators have observed in vivo (reduction of >50% of tumor growth) and hypothesize that metformin could be specifically efficient to treat up-front patients affected by OXPHOS+ GBM, in association with the standard first-line treatment with radiotherapy and temozolomide (RT-TMZ).

The investigators set up a dedicated molecular analysis including RNA assay and expression of OXPHOS markers for formalin-fixed paraffin-embedded tumors (FFPE), which allows to detect OXPHOS+ GBM at diagnosis.

Here a phase II, open label, non-randomized multicenter trial including five French neurooncology centers (H. Foch-Suresnes, Pitié-Salpêtrière-Paris, Saint Louis-Paris, Lyon, Marseille) and one in Italy (Istituto Besta, Milan) is proposed.

Newly diagnosed IDH wild-type GBM patients with the OXPHOS+ signature will be eligible for inclusion in this trial. The investigators expect to screen 640 patients and to include 64 patients over a period of 24 months with 24 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed informed consent for selection and treatment phase obtained from the patient/legal representative prior to performing any protocol-related procedures,
2. Patients must be willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits, and examinations including follow-up,
3. Newly-diagnosed histologically-confirmed supra-tentorial IDHwt glioblastoma (Grade 4 malignant glioma by World Health Organization, including gliosarcoma),
4. OXPHOS+ subtype by the central laboratory
5. No prior treatment for GBM other than surgery,
6. Substantial recovery from surgical resection, no major ongoing safety issues (eg, infection requiring I.V. antibiotics) following surgery,
7. Without corticosteroids or with stable dose of corticosteroids (ie ≤ dexamethasone 6 mg, methylprednisolone 30 mg or prednisone 38 mg),
8. ECOG (Eastern Cooperative Oncology Group) performance status 0-2,
9. Able to receive concomitant radio-chemotherapy according to the Stupp protocol (60Gy) based on investigator judgment,
10. Adequate bone marrow and normal hepatic function,
11. Creatinine clearance ≥ 30 mL/min (between 30 and 50 ml/min, patients will be prescribed no more than 1500mg of metformin),
12. Able to start RT within 7 weeks after histological diagnosis,
13. Patients must have life expectancy ≥ 16 weeks,
14. Patients affiliated to an appropriate health insurance system,
15. Age ≥ 18 years old,
16. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to the start of study drug,
17. Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception from the signing of the informed consent and continue throughout period of taking study treatment and for 30 days after last dose of study drug (duration of ovulatory cycle) plus the time required for the investigational drug to undergo five half-lives (both TMZ and metformin). The terminal half-life of temozolomide is 1.8 hours. The terminal half-life for metformin is 6.5 hours.
18. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception throughout the period of taking study treatment and for 6 months plus the time required for the investigational drug to undergo five half-lives (both TMZ and metformin). The terminal half-life of temozolomide is 1.8 hours. The terminal half-life for metformin is 6.5 hours.
19. White blood cells (WBC) ≥ 2000/μL
20. Neutrophils ≥ 1500/μL,
21. Platelets ≥ 100 x103/μL,
22. Hemoglobin ≥ 9.0 g/dL,
23. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 30 mL/min (using the Cockcroft-Gault formula) Female CrCl = (140-age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL Male CrCl = (140-age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL
24. Aspartate AminoTransferase (AST) ≤ 3.0 x ULN,
25. Alanine Aminotransferase (ALT) ≤ 3.0 x ULN,
26. Total Bilirubin ≤ 1.5 x ULN (except patients with Gilbert Syndrome who may have a total bilirubin < 3.0 x ULN).

Exclusion Criteria:

1. Prior treatment for GBM (other than surgical resection) including Gliadel wafer,
2. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years,
3. Any known metastatic extracranial or leptomeningeal disease,
4. IDH mutant,
5. Secondary GBM (ie, progression from prior low-grade or anaplastic glioma),
6. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the patient to receive protocol therapy, or interfere with the interpretation of study results,
7. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication (inflammatory bowel disease, major bowel resection),
8. Pregnant or breast-feeding women,
9. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV) and are receiving anti-viral therapy,
10. Patients with known active hepatitis (i.e., Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV)),
11. Patients with a known hypersensitivity to metformin and temozolomide or any of the excipients of the products,
12. Patients with severe renal insufficiency ie, CrCl < 30 mL/min (who should not receive contrast materials),
13. History or evidence upon physical/neurological examination of other central nervous system condition (eg, seizures, abscess) unrelated to cancer, unless adequately controlled by medication or considered not potentially interfering with protocol treatment,
14. Patients unable (eg, due to pacemaker or Implantable Cardioverter Defibrillator (ICD) device) or unwilling to have a contrast-enhanced MRI of the head,
15. Any acute medical condition that may impair renal function such as dehydration, severe infection, shock,
16. Any disease which may cause tissue hypoxia such as decompensated heart failure, respiratory failure, recent myocardial infarction
17. Past Diabetic precoma
18. Past Acute metabolic acidosis,
19. Alcohol intoxication and Alcoholism,
20. Persons protected by a legal regime (guardianship, trusteeship),
21. Prisoners or patients who are involuntarily incarcerated,
22. Patients who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Assessement of Progression Free Survival (PFS) of patients with newly-diagnosed IDH wild-type OXPHOS + GBM (either with or without FGFR3-TACC3 gene fusion) treated with RT plus TMZ combined with metformin | During the 24 months of follow-up
  Progression free survival (PFS) estimated by the RANO (Response Assesment in Neuro Oncology) criteria

SECONDARY OUTCOMES:
Assessement of the Overall survival (OS) of treated patients | During the 24 months of follow-up
  Overall survival (OS)
Assessement of the Overall Response rate (ORR) | During the 24 months of follow-up
  Overall response rate (ORR) estimated by the RANO criteria
Assessement of the the safety of metformin in association with concomitant RT-TMZ | During the 24 months of follow-up
  Type, frequency, and severity (grade III and IV toxicity) of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Assessement of the the tolerability of metformin in association with concomitant RT-TMZ | During the 24 months of follow-up
  Dose interruptions, reductions and dose intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Luisa DI STEFANO, MD, Principal Investigator — Foch Hospital
Locations (7):
- France (5):
  - Foch Hospital, Suresnes, Hauts de Seine
  - Hôpital Neurologique Pierre Wertheimer, Bron, Lyon
  - Timone Hospital, Marseille, Marseille
  - Saint Louis Hospital, Paris, Paris
  - Pitié Salpêtrière Hospital, Paris, PARIS
- Italy (2):
  - Istituto Nazionale Carlo Besta, Milan, Milano
  - Spidali Riuniti Di Livorno, Livorno, Toscana Nord Ouest

IPD SHARING:
Plan to Share IPD: No